CLINICAL TRIAL: NCT03262207
Title: Epigenetic Integrity of Spermatozoa in Patients With Germinal Testicular Tumours: Potential Risks and Consequences for the Conceptus
Brief Title: Epigenetic Integrity of Spermatozoa in Patients With Germinal Testicular Tumours
Acronym: GAMETH
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: DESCH AOI 2016
Record Dates: First submitted 2017-08-23; First posted 2017-08-25 (Actual); Last update posted 2017-08-25 (Actual); Status verified 2017-08

CONDITIONS: Seminomas
MeSH Terms: conditions — Seminoma | interventions — Flow Cytometry

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- testicular tumours
  Interventions: Other: Extraction genomic DNA; Other: Analysis of methylation profiles of numerous GSI and TE; Other: Analysis of methylation for the whole genome (sub-population of 15 samples from group 1); Other: Method of protein detection by immunostaining and flow cytometry
- fertile
  Interventions: Other: Extraction genomic DNA; Other: Analysis of methylation profiles of numerous GSI and TE; Other: Method of protein detection by immunostaining and flow cytometry
- infertile
  Interventions: Other: Extraction genomic DNA; Other: Analysis of methylation profiles of numerous GSI and TE; Other: Method of protein detection by immunostaining and flow cytometry

INTERVENTIONS:
Other: Extraction genomic DNA
Other: Analysis of methylation profiles of numerous GSI and TE
Other: Analysis of methylation for the whole genome (sub-population of 15 samples from group 1)
  Groups: testicular tumours
Other: Method of protein detection by immunostaining and flow cytometry

SUMMARY:
Recent data suggest that sperm cells carry an epigenetic message during spermatogenesis and that this message is crucial for the future development of the embryo. This epigenetic signature is notably represented by methylation of genes subjected to imprinting (GSI) and the methylation of transposable elements (TE). Data on the maintenance of the imprint and of the control of TE accompanying human gametogenesis in a context of adult germinal testicular cancers, seminomas, are extremely fragmentary for tumour tissues and inexistent for gametes.

The aim of this study is to determine whether patients with seminomas in comparison with fertile men carry a higher risk of presenting epigenetic alterations affecting their gametes.

This study is based on the use of an existing collection of biological samples. 90 samples will be selected and split into 3 groups:

* Group 1: 30 sperm samples from patients with seminomatous testicular tumours
* Group 2: 30 sperm samples from fertile patients
* Group 3: 30 sperm samples from infertile patients

After treatment of the samples (thawing, cell sorting and removal of cryoprotectants), they will be analysed.

ELIGIBILITY:
Inclusion Criteria:

* biological samples from persons who have provided written consent
* biological samples of patients over 18 years old
* with testicular tumours/Fertile/Infertile
* Matched for age with patients suffering from testicular tumours

Exclusion Criteria:

* biological samples of persons without national health insurance cover
* biological samples from patients with chronic hepatitis B or C or HIV infection

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: seminomas
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Analysis of methylation profiles in paternal genes subjected to imprinting (GSI) | at baseline

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France